CLINICAL TRIAL: NCT06637514
Title: A Phase 2 Study of JNT-517 in Adolescent Participants With Phenylketonuria
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JNT517-201
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- JNT-517 - 75 mg BID (Experimental): Drug: JNT-517 Tablet
  Interventions: Drug: JNT-517 Tablet
- Placebo - BID (Placebo Comparator): Drug: Placebo Tablet
  Interventions: Other: Placebo
- JNT-517 - 150 mg BID (Experimental): Drug: JNT-517 Tablet - 150 mg BID is a potential dose that may be used in the study. After safety, efficacy and pharmacokinetic data (PK) data have been reviewed for the first 5 participants assigned in the study, a decision will be made to increase dosage for additional participants.
  Interventions: Drug: JNT-517 Tablet

INTERVENTIONS:
Drug: JNT-517 Tablet — JNT-517: 75 mg BID
  Arms: JNT-517 - 75 mg BID
Other: Placebo — Placebo Tablet: BID
  Arms: Placebo - BID
Drug: JNT-517 Tablet — JNT-517: 150 mg BID
  Arms: JNT-517 - 150 mg BID

SUMMARY:
The goal of this Phase 2, randomized study is to assess the safety, tolerability, and pharmacokinetics (PK) of oral JNT-517 in adolescents (12 to less than 18 years of age) with PKU. Participants will receive either JNT-517 or placebo and will be blinded to their treatment assignment. Participants will have a 4 in 5 (or 80%) chance of receiving JNT-517. The study will last for up to 63 days including a Screening period, Treatment period and Follow-up period for safety.

Participants will:

* Take 75 mg JNT-517 or a placebo BID (2x per day) for 28 days
* Visit the clinic or have a mobile health nurse visit your home for checkups and tests
* Collect urine sample at home and bring to clinic on specified days
* Keep a food diary 3 days before each study visit

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females 12 to less than 18 years of age, inclusive on Day 1.
2. Clinical diagnosis of PKU.
3. Ability to swallow tablets.
4. Average of 2 plasma Phe levels during the Screening period greater than 360 μM and no plasma Phe level less than 300 μM.
5. Body weight equal or greater than 45 kg and body mass index less than 40 kg/m2.
6. Females of childbearing potential must practice sexual abstinence or agree to use 2 highly effective contraceptive methods.
7. Capable of giving signed informed consent (emancipated minors) or parent/legal guardian to provide informed consent and the participant to give assent and confirm ability to comply with study procedures.

Key Exclusion Criteria:

1. Any acute or chronic medical condition that would prevent the participant from complying with the procedures or place the participant at risk if they participate in the study.
2. Positive for hepatitis B or C or human immunodeficiency virus.
3. Any history of malignancy in the last 5 years, excluding nonmelanoma skin cancer.
4. Any history of liver disease.
5. Any history of cataracts or more than minimal cataracts observed during the Screening ophthalmologic examination.
6. Any surgical or medical conditions that may affect study drug absorption, distribution, metabolism, or excretion.
7. Creatinine clearance less than 90 mL/min by Cockcroft-Gault formula.
8. History of drug or alcohol abuse in the last year
9. Current, recent, or suspected infection within 14 days of Screening of SARS CoV 2/COVID 19.
10. Participation in another investigational drug trial within 30 days or, if known 5 half-lives of investigational drug (whichever is longer).
11. Unable to tolerate oral medication.
12. Allergy to JNT-517 or any component of the investigational product.
13. Received greater than 50 mL of blood or plasma within 30 days of Screening or greater than 500 mL of blood or plasma within 60 days of Screening.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Screening to Study Completion (Average of 9 weeks)
  Reported based on results of 12-lead electrocardiograms (ECGs), vital signs and clinical laboratory tests.

SECONDARY OUTCOMES:
Plasma AUC (area under the concentration-time curve) | Screening to Study Completion (Average of 9 weeks)
Cmax (maximum observed concentration) | Screening to Study Completion (Average of 9 weeks)
Tmax (time to Cmax) | Screening to Study Completion (Average of 9 weeks)
Change over time in plasma phenylalanine (Phe) and other amino acids | Screening to Study Completion (Average of 9 weeks)
Change over time in urinary phenylalanine (Phe) and other amino acids | Screening to Study Completion (Average of 9 weeks)

OTHER OUTCOMES:
Plasma metabolites of JNT-517 | Screening to Study Completion (Average of 9 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com